CLINICAL TRIAL: NCT06801119
Title: Dose-escalation Study to Assess the Safety, Tolerability, and Preliminary Efficacy of HN2301 in Patients with Relapsing and Refractory Systemic Lupus Erythematosus.
Brief Title: Efficacy and Safety of HN2301 in Refractory Systemic Lupus Erythematosus (SLE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen MagicRNA Biotechnology Co., Ltd (Industry)
Collaborators: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN2301-001
Record Dates: First submitted 2025-01-15; First posted 2025-01-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HN2301 treatment group (Experimental)
  Interventions: Drug: HN2301 injection

INTERVENTIONS:
Drug: HN2301 injection — Three dose groups were set up, starting from the low dose group and climbing to explore the safe and effective dose.

SUMMARY:
This is an investigator-initiated trial designed to evaluate the safety, and efficacy of HN2301 in Relapsing and refractory systemic lupus erythematosus

DETAILED DESCRIPTION:
This study is a prospective exploratory clinical trial in subjects with Relapsing and refractory systemic lupus erythematosus. The objective is to evaluate the safety, initial efficacy of HN2301injection in Relapsing and refractory systemic lupus erythematosus

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 69 (inclusive), of any gender, diagnosed with SLE according to the 2019 EULAR/ACR SLE diagnostic criteria;
2. A history of SLE for at least 6 months, having used a stable standard treatment regimen for at least 8 weeks, with the dosage stabilized for 2 weeks, yet the disease remains active or has relapsed; Standard treatment refers to the stable use of the following drugs alone or in combination: non-steroidal anti-inflammatory drugs (NSAIDs), antimalarials, corticosteroids; immunosuppressants including cyclophosphamide, methotrexate, azathioprine, mycophenolate mofetil, leflunomide, tacrolimus, cyclosporine, etc.; targeted drugs include belimumab, rituxima, eculizumab, rituximab, etc.
3. Oral corticosteroids are prednisone (or equivalent drug) ≥7.5mg/day and ≤30mg/day. If used in combination with immunosuppressants, there is no minimum daily dose requirement;
4. At least two immunosuppressants have been used in a standardized manner (including hydroxychloroquine);
5. Screening period tests meet: positive blood antinuclear antibody (ANA), and/or positive anti-ds-DNA antibodies, and/or hypocomplementemia;
6. Screening period SLEDAI-2K score ≥6 points. If scoring includes low complement and/or anti-ds-DNA antibodies, the score for SLEDAI-2K clinical symptoms (excluding low complement and/or anti-ds-DNA antibodies) should be ≥4 points;
7. Appropriate bone marrow, coagulation, cardiopulmonary, liver, and kidney functions. Bone marrow function: ANC ≥1.5×10^9/L, ALC ≥0.8×10^9/L, Hb ≥80g/L. No use of transfusions and growth factors allowed within 7 days prior to screening to meet these requirements. Coagulation function: INR or APTT ≤1.5×ULN. Cardiac function: Echocardiography (ECHO) assessment of left ventricular ejection fraction (LVEF) ≥40%. Lung function: ≤CTCAE grade 1 dyspnea and SpO2 ≥92% (measured by pulse oximetry) while breathing indoor air. Liver function: ALT and AST ≤2.5×ULN, total bilirubin <2.0mg/dL (Gilbert syndrome subjects total bilirubin <3.0mg/dL). Kidney function: defined as creatinine clearance rate (Cockcroft-Gault) ≥50mL/min without need for fluid assistance;
8. Non-pregnant/non-lactating participants, willing to adopt contraceptive measures within 12 months after drug infusion.

Exclusion Criteria:

1. Individuals with positive Hepatitis B surface antigen (HBsAg) and/or Hepatitis B core antibody (HBcAb), and Hepatitis B virus (HBV) DNA positivity or titers above the detection threshold; those with positive Hepatitis C virus (HCV) antibodies and HCV RNA positivity or titers above the detection threshold; individuals with Human Immunodeficiency Virus (HIV) antibodies positivity, CMV DNA positivity or above the detection limit; those with positive syphilis antigen or antibodies;
2. Presence of other uncontrolled active infections;
3. History of major organ transplantation (such as heart, lung, liver, kidney) or bone marrow/hematopoietic stem cell transplantation;
4. Pregnant or breastfeeding women;
5. Receiving any mRNA-LNP product or other LNP medications within the past two years;
6. History of any of the following cardiovascular diseases within the last 6 months before screening: Class III or IV heart failure defined by the New York Heart Association (NYHA), myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias, or other clinically significant cardiac diseases;
7. History of live vaccine administration within the last 30 days;
8. Individuals with asthma, severe allergies;
9. Other conditions deemed inappropriate for participation in this clinical study by the investigator.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-03-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to HN2301 | 3 months
  Incidence and severity of AEs associated with HN2301 as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
vivo CAR T cell production | Day-28 to14 days
  CAR T production in the peripheral blood of systemic lupus erythematosus (SLE) patients, by flow cytometry (FACS), and quantitative polymerase chain reaction (qPCR) in peripheral blood
B cell ratio and counts in peripheral blood | Day-28 to12 months
  Assessment of B cell ratio and counts (B cell counts per μl peripheral blood) and B cell subsets(naive B cell, memory B cell) by flow cytometry (FACS) in peripheral blood
Change from baseline of SLEDAI-2K score after HN2301 administration. | Day-28 to12 months
  Assessment of Systemic Lupus Erythematosus Disease Activity Index 2000 from baseline administration at various timepoints up to month 12 follow-up visit. A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
Quantify the clinical activity of HN2301 in patients with SLE using Physician Global Assessment (PGA) . | Day-28 to12 months
  Assessment of Physician Global Assessment (PGA) from baseline administration at various timepoints up to month 12 follow up visit. A total score can fall between 0.0 and 3.0, with a higher score representing a more significant degree of disease activity.
Proportion of patients achieving low disease activity status (LLDAS) after HN2301 administration | Day-28 to12 months
  Assessment of LLDAS maintenance rate at various timepoints up to the month 12 follow-up visit.
Proportion of patients achieving DORIS remission after HN2301 administration | Day-28 to12 months
  Assessment of DORIS response rate at various timepoints up to the month 12 follow-up visit.
Assess the clinical activity of HN2301 in patients with SLE using Systemic Lupus Erythematosus Responder Index-4 (SRI-4) | Day-28 to12 months
  Assessment of whether participants meet the Systemic Lupus Erythematosus Responder Index-4 (SRI-4) criteria (yes/no) at various timepoints up to the month 12 follow-up visit.
Proportion of patients achieving complete renal response (CRR) after HN2301 administration | Day-28 to12 months
  Proportion of patients achieving complete renal response (CRR) after HN2301 administration

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Chen, MD, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided